CLINICAL TRIAL: NCT05781399
Title: A Phase 1/2, First-In-Human, Multiple Part, Single Ascending and Multiple Dose Study of JNT-517 in Healthy Participants and in Participants With Phenylketonuria
Brief Title: First-in-Human, Multiple Part Clinical Study of JNT-517 in Healthy Participants and in Participants With Phenylketonuria
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JNT517-101
Record Dates: First submitted 2023-02-11; First posted 2023-03-23 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Phenylketonuria
Keywords: PKU
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Intervention Model Description: The study will be conducted in 6 parts: Parts A, B, C,D, E, and F. This study will be seamless, meaning various study parts could begin while other parts are still ongoing, but dose escalation will occur only after satisfactory review of safety and tolerability data from a minimum of 6 participants completing through Day 3, and available PK data.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Parts A, B, D, and F are blinded. Parts C and E are open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- JNT-517 SAD (Part A and Part F) (Experimental): Single dose of JNT-517 or placebo in fasted state.
  Interventions: Drug: JNT-517 Suspension; Drug: Placebo Suspension
- JNT-517 MAD (Part B) (Experimental): JNT-517 or placebo once or twice daily for 14 days, with first daily dose given after an overnight fast.
  Interventions: Drug: JNT-517 Suspension; Drug: Placebo Suspension
- JNT-517 Suspension Then Tablet Fasted Then Tablet Fed (Part C) (Experimental): Single dose of JNT-517 suspension, JNT-517 tablet in a fasted state, and JNT-517 tablet in a fed state in a sequential, open-label manner. Each treatment is separated by a minimum of 5 half-lives.
  Interventions: Drug: JNT-517 Suspension; Drug: JNT-517 Tablet
- JNT-517 Tablet Fasted Then Tablet Fed Then Suspension (Part C) (Experimental): Single dose of JNT-517 tablet in a fasted state, JNT-517 tablet in a fed state, and JNT-517 suspension in a sequential, open-label manner. Each treatment is separated by a minimum of 5 half-lives.
  Interventions: Drug: JNT-517 Suspension; Drug: JNT-517 Tablet
- JNT-517 Tablet Fed Then Suspension Then Tablet Fasted (Part C) (Experimental): Single dose of JNT-517 tablet in a fed state, JNT-517 suspension, and JNT-517 tablet in a fasted state in a sequential, open-label manner. Each treatment is separated by a minimum of 5 half-lives.
  Interventions: Drug: JNT-517 Suspension; Drug: JNT-517 Tablet
- JNT-517 PKU (Part D and E) (Experimental): JNT-517 or placebo daily for 4 weeks. Dose is based on data from Parts A, B, and C.
  Interventions: Drug: JNT-517 Tablet; Drug: Placebo Tablet

INTERVENTIONS:
Drug: JNT-517 Suspension — JNT-517 in on-site compounded suspension
  Arms: JNT-517 MAD (Part B); JNT-517 SAD (Part A and Part F); JNT-517 Suspension Then Tablet Fasted Then Tablet Fed (Part C); JNT-517 Tablet Fasted Then Tablet Fed Then Suspension (Part C); JNT-517 Tablet Fed Then Suspension Then Tablet Fasted (Part C)
Drug: Placebo Suspension — On-site compounded placebo suspension
  Arms: JNT-517 MAD (Part B); JNT-517 SAD (Part A and Part F)
Drug: JNT-517 Tablet — JNT-517 tablets, 25 mg and 75 mg
  Arms: JNT-517 PKU (Part D and E); JNT-517 Suspension Then Tablet Fasted Then Tablet Fed (Part C); JNT-517 Tablet Fasted Then Tablet Fed Then Suspension (Part C); JNT-517 Tablet Fed Then Suspension Then Tablet Fasted (Part C)
Drug: Placebo Tablet — Matching film-coated placebo tablet
  Arms: JNT-517 PKU (Part D and E)

SUMMARY:
The goal of Parts A and B of this Phase 1/2, first-in-human, randomized study is to assess the safety, tolerability, and pharmacokinetics (PK) of single (SAD) and multiple (MAD) ascending doses of oral JNT-517 in healthy participants. In Part C, the goal is to evaluate the differences in bioavailability between a tablet and suspension formulation of JNT-517 and the food effect in healthy volunteers. All participants in Part C will receive JNT-517. The goal of Part D is to assess the safety, tolerability, PK, and effect on urinary Phe and other amino acids of JNT-517 in participants with phenylketonuria (PKU). Participants in Part D will receive either JNT-517 or placebo and will be blinded to their treatment assignment.

The study consists of 6 parts:

* Part A: SAD in healthy participants -randomized, double-blind, placebo-controlled
* Part B: MAD in healthy participants (14 days)-randomized, double-blind, placebo-controlled
* Part C: Relative bioavailability of 2 formulations and food effect in healthy participants-randomized, open-label
* Part D: Phase 2 in participants with PKU (4 weeks)-randomized, double-blind, placebo-controlled
* Part E: Phase 2 in participants with PKU (4 weeks) open label
* Part F: SAD Phase 1 in healthy participants, randomized, double-blind, placebo-controlled

In each part, participants will complete a Screening Period, a Treatment Period, and a Follow-up Period for safety.

ELIGIBILITY:
Key Inclusion Criteria:

Parts A, B, C, and F:

1. Males and females 18 to 55 years of age.
2. Medically healthy with no clinically significant medical history.
3. Body mass index (BMI) of 18-40 kg/m2 and total body weight >50 kg (110 lbs).
4. Non-smoker for at least 2 weeks prior to dosing and willing to abstain during the study.

   Part D and E:
5. Males and females 18 to 65 years of age, inclusive.
6. Diagnosis of PKU with a confirmed genotype.
7. At least 2 plasma Phe levels >600 μM over the past 12 months.
8. BMI of 18-40 kg/m2.

   All Parts:
9. Females of childbearing potential must agree to use 2 highly effective contraceptive methods.
10. Capable of giving signed informed consent and able to comply with study procedures.

Key Exclusion Criteria:

All Parts:

1. Any acute or chronic medical condition that would prevent the participant from complying with the procedures or place the participant at risk if they participate in the study.
2. Positive for hepatitis B or C or human immunodeficiency virus.
3. Any history of malignancy in the last 5 years, excluding non-melanoma skin cancer.
4. Any history of liver disease.
5. Any surgical or medical conditions that may affect study drug absorption, distribution, metabolism, or excretion.
6. Participation in another investigational drug trial within 30 days or, if known, 5 half-lives of the investigational drug (whichever is longer).
7. History of drug/alcohol abuse in the last year.
8. Current, recent, or suspected infection within 4 weeks of Screening of SARS-CoV-2/COVID-19.
9. Received a vaccine for SARS-CoV-2/COVID-19 within 14 days of Screening.
10. Unable to tolerate oral medication.
11. Allergy to JNT-517 or any component of the investigational product.
12. Received >50 mL of blood or plasma within 30 days of Screening or >500 mL of blood or plasma within 60 days of Screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events | Parts A/C/F: Screening to Day 8; Part B: Screening to Day 21; Part D/E: Screening to Day 35
  Reported based on results of 12-lead ECGs, vital signs, clinical laboratory tests, and other medical assessments.

SECONDARY OUTCOMES:
Plasma area under the concentration-time curve (AUC) of JNT-517 | Parts A/C/F: pre-dose to 72 hrs post-dose on Day 1; Part B: pre-dose to 24 hrs post-dose on Days 1, 14 and pre-dose on Days 3, 13; Part D/E: pre-dose to 4 hrs post-dose on Days 1, 14, 28
Maximum observed plasma concentration (Cmax) of JNT-517 | Parts A/C/F: pre-dose to 72 hrs post-dose on Day 1; Part B: pre-dose to 24 hrs post-dose on Days 1, 14 and pre-dose on Days 3, 13; Part D/E: pre-dose to 4 hrs post-dose on Days 1, 14, 28
Time to maximum plasma concentration (Tmax) of JNT-517 | Parts A/C/F: pre-dose to 72 hrs post-dose on Day 1; Part B: pre-dose to 24 hrs post-dose on Days 1, 14 and pre-dose on Days 3, 13; Part D/E: pre-dose to 4 hrs post-dose on Days 1, 14, 28
Plasma terminal half-life (t1/2) of JNT-517 | Parts A/C/F: pre-dose to 72 hrs post-dose on Day 1; Part B: pre-dose to 24 hrs post-dose on Days 1, 14 and pre-dose on Days 3, 13; Part D/E: pre-dose to 4 hrs post-dose on Days 1, 14, 28
Comparison of Tmax of JNT-517 in fed and fasted states | Pre-dose to 72 hrs post-dose on Day 1
  Part C only
Comparison of Cmax of JNT-517 in fed and fasted states | Pre-dose to 72 hrs post-dose on Day 1
  Part C only
Comparison of AUC of JNT-517 in fed and fasted states | Pre-dose to 72 hrs post-dose on Day 1
  Part C only
Changes in urinary amino acid levels | Screening and Days 1, 7, 14, 21, 28
  Part D/E only. Urine samples will be collected at the indicated timepoints and analyzed for amino acid levels, including Phe.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (11):
  - University of Florida College of Medicine, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - Rare Disease Research, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Oregon Health & Sciences University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Utah Health - The University of Utah Hospital, Salt Lake City, Utah
- Australia (4):
  - Nucleus Network Melbourne, Melbourne, Melbourne VIC
  - Westmead Hospital, Westmead, New South Wales
  - Mater Misericordia Ltd, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com